CLINICAL TRIAL: NCT00304291
Title: A Pilot Study of Mitoxantrone for the Treatment of Recurrent Neuromyelitis Optica (Devic's Disease)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Principal Investigator, Bianca Weinstock-Guttman, Principal Investigator, State University of New York at Buffalo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JNI-NMO-101
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Neuromyelitis Optica; Myelitis, Transverse; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases of the Nervous System
Keywords: Novantrone
MeSH Terms: conditions — Neuromyelitis Optica; Myelitis, Transverse; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases of the Nervous System | interventions — Mitoxantrone

INTERVENTIONS:
Drug: Mitoxantrone

SUMMARY:
Neuromyelitis optica (NMO) is a severe demyelinating disease that selectively involves the optic nerves and the spinal cord but usually spares the brain. NMO is considered to have a B cell induced pathogenesis. Mitoxantrone (MITO, Novantrone®), a synthetic anthracenedione approved for worsening relapsing-remitting multiple sclerosis (MS) and secondary progressive MS, has been shown to primarily suppress the humoral response. We conducted a prospective 2-year study to evaluate the benefit of MITO in five relapsing NMO patients.

DETAILED DESCRIPTION:
The treatment protocol consisted of monthly 12 mg/m2 MITO intravenous infusions for 6 months followed by 3 additional treatments every 3 months. Neurological assessment including the determination of the Expanded Disability Status Scale (EDSS) score was performed every 3 months and during relapses. Orbital, brain and spinal cord MRI was performed at baseline, 3, 6, 12, 18, and 24 months. Visual evoked potentials and ophthalmologic evaluations were performed at baseline and annually.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent longitudinal myelitis (>3 segments of spinal cord involvement by MRI) with or without recurrent ON (unilateral or bilateral) but with normal brain MRI.
* Patients with recurrent longitudinally extensive myelitis without optic neuritis have an underlying pathology and serology similar to NMO and it is appropriate to consider this a form of NMO10.
* Cerebrospinal fluid required no intrathecal IgG synthesis or oligoclonal bands.
* Age was required to be 18-55 years
* Extended Disability Status Score ≤ 7.

Exclusion Criteria:

* Cardiac risk factors (e.g history of congestive heart failure and left ventricular ejection fraction (LVEF) < 50%
* Systemic diseases such as lupus, Sjogren's syndrome, anti-phospholipid antibody syndrome, sarcoidosis, rheumatoid arthritis, or vitamin B12 deficiency
* Previous treatment with mitoxantrone or anthracyclines

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5
Dates: Start 2001-08; Study Completion 2004-05

PRIMARY OUTCOMES:
Relapse rate

SECONDARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Weinstock-Guttman, M.D., Study Director — Baird Multiple Sclerosis Center
Locations (1):
- Baird Multiple Sclerosis Center, Buffalo, New York, United States

REFERENCES:
- [Result] Weinstock-Guttman B, Ramanathan M, Lincoff N, Napoli SQ, Sharma J, Feichter J, Bakshi R. Study of mitoxantrone for the treatment of recurrent neuromyelitis optica (Devic disease). Arch Neurol. 2006 Jul;63(7):957-63. doi: 10.1001/archneur.63.7.957. PMID 16831964